CLINICAL TRIAL: NCT05207202
Title: Effect of EIT-guided PEEP Titration on the Prognosis of Patients with Moderate to Severe ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Director of Intensive Care Unit, Principal Investigator, Clinical Professor, Southeast University, China
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021010065
Record Dates: First submitted 2021-12-15; First posted 2022-01-26 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Clinical Outcomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EIT-PEEP strategy (Active Comparator): Patients will receive PEEP titrated by EIT with a stepwise decrease PEEP trial
  Interventions: Device: electrical impedance tomography
- ARDSNet-PEEP strategy (Active Comparator): PEEP will be set according to the low FiO2-PEEP table to keep the oxygenation goals: SpO2 between 88% and 95%, and PaO2 between 55mmHg and 80mmHg.
  Interventions: Device: electrical impedance tomography

INTERVENTIONS:
Device: electrical impedance tomography — PEEP titrated by EIT will be performed with a decremental trial at the enrollment. Right after completing RM, PEEP will be set to 20cmH2O and then reduced in steps of 2cmH2O from 20 to zero every 2min.

SUMMARY:
Acute respiratory syndrome distress (ARDS) is a clinical common syndrome with high mortality. Mechanical ventilation (MV) is the cornerstone of management of ARDS but can lead to ventilator-induced lung injury. Positive end-expiratory pressure (PEEP), as one of main component of MV, has been widely used in the clinical practice. However, the PEEP selection is still a difficult problem for moderate to severe ARDS patients. EIT, an imaging tool evaluating the regional ventilation distribution at the bedside, can achieve the individual PEEP selection for all mechanically ventilated patients. This article compared the effect of PEEP titrated guided by EIT with fraction of inspired oxygen (FiO2)-PEEP table on the clinical outcomes.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-blind, parallel-group, adaptive randomized controlled trial (RCT) with intention-to-treat analysis which aims to determine the effects of PEEP setting guided by EIT on the clinical outcomes for moderate or severe ARDS patients ventilated with lung protective ventilation strategy. Adult patients with moderate to severe ARDS less than 72 hours after diagnosis will be included in this study. Patients in the intervention group will receive PEEP titrated by EIT with a stepwise decrease PEEP trial, whereas patients in the control group will select PEEP based on the FiO2-PEEP table. Other ventilator parameters will be set according to the ARDSnet strategy. The primary outcome is 28-day mortality. The secondary outcomes include ventilator-free days and shock-free days at day 28, length of ICU and hospital stay, the rate of successful weaning, proportion requiring rescue therapies, compilations, respiratory variables, and Sequential Organ Failure Assessment (SOFA). This study will also perform the interim analysis and subgroup analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years
2. Moderate-to-severe ARDS, defined by the ARDS Definition Task Force in the Berlin definition (partial pressure of arterial oxygen [PaO2]:FiO2 ratio ≤200 mmHg with a PEEP ≥5 cmH2O)
3. Diagnosis of ARDS less than 72 hours

Exclusion Criteria:

1. Expected to be mechanically ventilated for less than 48 hours
2. Severe chronic respiratory diseases requiring long-term home oxygen therapy or noninvasive MV
3. Undrained pneumothorax or subcutaneous emphysema
4. Undergoing extracorporeal membrane oxygenation (ECMO) before enrollment
5. Contraindication to the use of EIT (pacemaker, automatic implantable cardioverter defibrillator, and implantable pumps)
6. Severe neuromuscular disease
7. Hemodynamic instability
8. Contraindications to hypercapnia, such as intracranial hypertension or acute coronary syndrome
9. Severe other organs dysfunction with a low expected survival (7 days) or palliative care
10. Solid organ or hematologic tumors with the expected survival time less than 30 days
11. Participating in other clinical trials within 30 days
12. Pregnancy
13. Refusal to sign the informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
28-day mortality | at day 28
  mortality in Day 28

SECONDARY OUTCOMES:
VFDs at day 28 | at day 28
  defined as the number of days between successful weaning from MV and day 28 after study enrollment
Shock-free days at day 28 | at day 28
  Shock-free days at day 28
Length of ICU stay | up to 24 months
  the survival rate(survival/total) during ICU stay
Length of hospital stay | up to 24 months
  the survival rate(survival/total) during hospital stay
The rate of successful weaning | at day 28
  Proportion of people who are not dependent on ventilator ventilation
Proportion requiring rescue therapies | day 28
  Proportion of people who require rescue therapies
Rate of pneumothorax | day 28
  Rate of pneumothorax
driving pressure | day 0, day 1, day 2, day 3, day 7
  measurement as one index of respiratory compliance at day 0, 1, 2, 3, and 7 from enrollment
Sequential Organ Failure Assessment (SOFA) score at the time of enrollment | at the time of enrollment
  SOFA range from three to eight. The higher the score, the worse the prognosis
Blood pressure at day D1, 2, 3, and 7 from enrollment | up to 24 months
  Both systolic and diastolic pressure at day D1, 2, 3, and 7 from enrollment
respiratory rate | up to 7 days
  respiratory rate
number of shock and gastrointestinal hemorrhage | day 28
  shock, and gastrointestinal hemorrhage

OTHER OUTCOMES:
blood gas | 28 day
  blood gas and the change at each time point
vital signs | 28 day
  HR, MAP, RR, SPO2, CVP, CO and so on at each time point
Ventilator parameters and respiratory mechanics | 28 day
  VT, RR, PEEP, FiO2, compliance, resistance and so on

CONTACTS AND LOCATIONS:
Overall Officials: ling liu, phD, Study Director — Southeast University, China
Locations (5):
- China (5):
  - the First Affiliated Hospital of Guangzhou Medical University, Department of Critical Care Medicine, Guangzhou, Guangdong
  - Department of Critical Care Medicine, Zhongda Hospital, School of Medicine, Southeast University, Nanjing, Jiangsu
  - Department of Critical Care Medicine, Renji Hospital, Shanghai, Shanghai Municipality
  - Department of Critical Care Medicine, Zhongshan Hospital of Fudan University, Shangha, Shangha
  - Department of ICU, Sichuan Academy of Medical Sciences and Sichuan Provincial People's Hospital, Chengdu, Sichuan

REFERENCES:
- [Derived] Yuan X, Zhang R, Wang Y, Chen D, Chao Y, Xu J, Guo L, Liu A, Xie J, Pan C, Yang Y, Qiu H, Liu L. Effect of EIT-guided PEEP titration on prognosis of patients with moderate to severe ARDS: study protocol for a multicenter randomized controlled trial. Trials. 2023 Apr 11;24(1):266. doi: 10.1186/s13063-023-07280-6. PMID 37041561